CLINICAL TRIAL: NCT04642534
Title: Molecular and Functional Interplay Between the Circadian Clocks and Eating Patterns in Patients with Cardio-metabolic Diseases (Cohort)
Brief Title: Circadian Clocks and Eating Patterns (Cohort)
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Jardena Puder, Principal investigator, University of Lausanne Hospitals
Other Study IDs: 2019-01207
Record Dates: First submitted 2020-11-02; First posted 2020-11-24 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2022-10

CONDITIONS: Postpartum Women; Diabetes, Gestational
Keywords: Circadian rhythms; Metabolic syndrome; Eating duration; Sleep/wake cycles
MeSH Terms: conditions — Diabetes, Gestational; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Blood, serum and plasma Skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Postpartum women who had gestational diabetes mellitus: Inclusion at 4-8 weeks postpartum Follow-up for 6 months
- Postpartum women after an uneventful pregnancy: Inclusion at 4-8 weeks postpartum Follow-up for 6 months

SUMMARY:
For women of reproductive age, the overall postpartum weight retention (weight gain between pregnancies) plays a significant role in long-term obesity. With 20% of women retaining ≥ 5 kg at 12 months postpartum, the risk of developing conditions, such as gestational diabetes mellitus (GDM), metabolic syndrome (MS) and subsequently diabetes and cardiovascular diseases, is substantially increased. In post-GDM mothers (women who had GDM in their recent pregnancy), postpartum weight retention is also an essential predictor of future diabetes.

Recent studies have identified the impact of circadian rhythms (influencing sleep/wake cycles) and diurnal rhythm of eating (when and how often calories are consumed over a 24h period) on cardio-metabolic disorders. In women, one remarkable feature of the postpartum period is an 'externally imposed' circadian misalignment of both sleep and eating rhythms, because most babies take several weeks to months to establish their daily pattern of activity and feeding, which is particularly relevant for breastfeeding women, as the responsibility is generally on the mother.

The overarching goal of this project is to explore the interplay between the diurnal rhythm of eating, circadian and metabolic parameters in humans. The potential postpartum effects of circadian disruption will be unraveled in women who had GDM during their pregnancy and those with an uneventful pregnancy. These women are subject to a circadian misalignment due to their 'externally imposed' changes in sleep/wake cycles and eating times in the postpartum period.

With a comprehensive approach combining molecular characterization of in vivo and in vitro circadian clock parameters along with metabolic, endocrine, transcriptomic, and lipidomic studies, the investigators will assess if eating duration and/or circadian misalignment impact on circadian clock parameters of postpartum women in a prospective cohort of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Breastfeeding mothers at 4-8 week postpartum
* With or without gestational diabetes mellitus diagnosed at 24-32 gestational weeks, according to the International Association of Diabetes and Pregnancy Study Groups (IADPSG) consensus criteria
* Confident use of a smartphone and able to take regular pictures of food/drinks

Exclusion Criteria:

* Pre-existing diabetes (prior to pregnancy)
* Major illness/fever over the 2 weeks (prior to the visits with blood tests)
* Shift work or work at irregular hours planned after maternity leave
* Active cancer and/or oncologic treatment over the previous 12 months
* Coagulation disorder, on regular anticoagulant drug, skin disorder affecting wound healing
* Enrolled in a clinical trial / intervention study
* Major known mental illness, unable to give informed consent
* Inability to follow the study procedures

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Postpartum women followed at the Lausanne University Hospital (CHUV)
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Eating duration | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Duration from the first to last caloric intake over 24-hour cycle
Correlation of in vitro circadian parameters (amplitude and magnitude) with clinical metabolic health outcomes (body weight) | At baseline
  Measured in cultured skin fibroblasts

SECONDARY OUTCOMES:
Sleep/wake cycles | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Measured by actigraphy
Sleep/wake cycles | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Measured by the Pittsburgh Sleep Quality Index (scale 0-21, 0 indicating no sleeping difficulty, 21 indicating severe sleeping difficulties)
Body weight | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Measured by bioelectrical impedance analysis
Fat mass | Changes between baseline and the close-out visit (i.e.changes between Month 0 and Month 6)
  Measured by bioelectrical impedance analysis
Fat-free mass | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Measured by bioelectrical impedance analysis
Physical activity (activity count per minute) | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Measured by actigraphy
Fasting glucose | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Measured by clinical chemistry
Lipid profile (concentration of total cholesterol, LDL cholesterol, triglycerides, HDL cholesterol) | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Measured by clinical chemistry
Glucose excursion (time-in-range, coefficient of variation) | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Measured by continuous glucose monitoring

OTHER OUTCOMES:
Blood hormonal profile | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Insulin and thyroid-stimulating hormone (mIU/L)
Blood hormonal profile | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Cortisol (nmol/L)
Markers of lipid metabolism | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Measured by high-throughput mass spectrometry lipidomics
Metabolomic parameters of energy metabolism | Changes between baseline and the close-out visit (i.e. changes between Month 0 and Month 6)
  Measured by high-throughput mass spectrometry metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Jardena Puder, MD, Principal Investigator — University of Lausanne Hospitals; Tinh-Hai Collet, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Lausanne University Hospital (CHUV), Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips NE, Mareschal J, Biancolin AD, Sinturel F, Umwali S, Blanc S, Hemmer A, Naef F, Salathe M, Dibner C, Puder JJ, Collet TH. The metabolic and circadian signatures of gestational diabetes in the postpartum period characterised using multiple wearable devices. Diabetologia. 2025 Feb;68(2):419-432. doi: 10.1007/s00125-024-06318-x. Epub 2024 Nov 12. PMID 39531039